CLINICAL TRIAL: NCT01932463
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound for Unilateral Thalamotomy in the Treatment of Tremor
Brief Title: ExAblate (Magnetic Resonance-guided Focused Ultrasound Surgery) for Treatment of Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD002
Record Dates: First submitted 2013-08-22; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Tremor; Essential Tremor
Keywords: Tremor; Essential Tremor; Medication-refractory Essential Tremor
MeSH Terms: conditions — Tremor; Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAb;ate MRgFUS (Experimental)
  Interventions: Device: ExAblate Transcranial System

INTERVENTIONS:
Device: ExAblate Transcranial System — MR Guided Focused Ultrasound
  Other Names: MRgFUS; FUS; Focused Ultrasound; MR Guided Focused Ultrasound

SUMMARY:
A feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound for Unilateral Thalamotomy in the Treatment of Tremor

DETAILED DESCRIPTION:
The non-invasive high-intensity focused ultrasound has been coupled with high resolution MRI to provide precise, consistent treatments that can be monitored in real-time. The development of phased array transducers allows for tightly focused treatment volumes and for the ability to compensate for distortions by tissue inhomogeneities. The landmark advance in MRgFUS for neurosurgeons occurred as the ability to sonicate through the intact cranium was achieved with phased array transducers and acoustic modeling using CT reconstructions of the skull. By coupling HIFU with MRI, detailed treatment plans can be generated and intra-procedure real-time monitoring is available. Standard MR sequences have been shown to reliably predict tissue damage during thermal lesioning with ultrasound. The precision of the technology has already been demonstrated in animal models and is currently being investigated in humans with brain tumors and neuropathic pain syndromes. Unlike stereotactic radiosurgery, the treatment can be monitored continuously in real time with MRI and MR-thermography. We anticipate that a MRgFUS non-invasive thermal lesioning is similarly as safe as DBS (or other current procedure and will provide several years of benefit through reduction of contralateral motor symptoms and potential medication side effects in ET, while still permitting subsequent treatment with DBS should that become clinically desirable.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, between 18 and 80 years, inclusive
2. Patients who are able and willing to give consent and able to attend all study visits
3. A diagnosis of ET as confirmed from clinical history and examination by a movement disorder neurologist
4. Tremor refractory to adequate trials of at least two medications, one of which should be either propranolol or primidone. An adequate medication trial is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated.
5. Vim nucleus of thalamus can be target by the ExAblate device. The Vim region of the thalamus must be apparent on MRI such that targeting can be performed with either direct visualization or by measurement from a line connecting the anterior and posterior commissures of the brain.
6. Able to communicate sensations during the ExAblate MRgFUS treatment
7. Postural or intention tremor severity score of greater than or equal to 2 in the dominant hand/arm as measured by the CRST rating scale.
8. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
9. May have bilateral appendicular tremor
10. Significant disability due to essential tremor despite medical treatment (CRST score of 2 or above in any one of the items 16-23 from the Disability subsection of the CRST: [speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working, and social activities])
11. Inclusion and exclusion criteria have been agreed upon by two members of the medical team.

Exclusion Criteria:

1. Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication
   * Patients with documented myocardial infarction within six months of protocol entry
   * Congestive heart failure requiring medication (other than diuretic)
   * Patients on anti-arrhythmic drugs
2. Alcohol or drug abuse within the past 6 months
3. Severe hypertension (diastolic BP > 100 on medication)
4. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
5. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
6. Severely impaired renal function (estimated glomerular filtration rate < 30ml/min/1.73 m2) or receiving dialysis
7. History of abnormal bleeding and/or coagulopathy
8. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
9. Active or suspected acute or chronic uncontrolled infection
10. History of intracranial hemorrhage
11. Cerebrovascular disease (multiple CVA or CVA within 6 months)
12. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
13. Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema)
14. Untreated, uncontrolled sleep apnea
15. Are participating or have participated in another clinical trial in the last 30 days
16. Patients unable to communicate with the investigator and staff.
17. Presence of any other neurodegenerative disease like parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease. The presence of some mild parkinsonian features will be accepted since ET is recognized to be associated with overlap symptoms of PD. The mild PD symptoms that will be tolerated for inclusion into the trial include resting tremor, bradykinesia, and rigidity.
18. Presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
19. History of immunocompromise, including patient who is HIV positive
20. Known life-threatening systemic disease
21. Patients with a history of seizures within the past year
22. Patients with psychiatric illness that are not well controlled. Any presence of psychosis will be excluded. Patients with mood disorders including depression will be excluded if they have exhibited symptoms within 6 months while on medication. Patients who have been treated with transcranial magnetic stimulation or ECT will be excluded.
23. Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter, PT > 14, PTT > 36 or INR > 1.3) or a documented coagulopathy
24. Patients with brain tumors
25. Any illness that in the investigator's opinion preclude participation in this study.
26. Pregnancy or lactation.
27. Legal incapacity or limited legal capacity.
28. Patients who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of Thalamotomy lesion | 1 day
  Comparison of the stereotactic coordinates of the atlas to the lesion created in the brain.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Yamamoto K, Sarica C, Elias GJB, Boutet A, Germann J, Loh A, Joel SE, Bigioni L, Gwun D, Gramer R, Li SX, Zemmar A, Vetkas A, Algarni M, Devenyi G, Chakravarty M, Hynynen K, Scantlebury N, Schwartz ML, Lozano AM, Fasano A. Ipsilateral and axial tremor response to focused ultrasound thalamotomy for essential tremor: clinical outcomes and probabilistic mapping. J Neurol Neurosurg Psychiatry. 2022 Aug 22:jnnp-2021-328459. doi: 10.1136/jnnp-2021-328459. Online ahead of print. PMID 35995551